CLINICAL TRIAL: NCT02249039
Title: Intravenous Clonidine for Sedation in Infants and Children Who Are Mechanically Ventilated - Dosing Finding Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00109563
Record Dates: First submitted 2014-08-11; First posted 2014-09-25 (Estimated); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Mechanical Ventilation Complication
MeSH Terms: interventions — Clonidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- intermittent IV CLON (Experimental): Mechanically ventilated infants and children receive intravenous intermittentClonidine
  Interventions: Drug: intermittent IV CLON

INTERVENTIONS:
Drug: intermittent IV CLON — Mechanically ventilated infants and children receive intravenous intermittent Clonidine instead of dexmedetomidine
  Other Names: clonidine hydrochloride; Duraclon

SUMMARY:
Critically ill infants and children who are mechanically ventilated are often given large doses of opiates and benzodiazepines to provide analgesia-sedation. These drugs significantly cause tolerance and dependence, depresses the drive to breathe, and thus prolongs the need for mechanical ventilation and the associated complications. We propose IV CLON could be used as effectively as DEX.

DETAILED DESCRIPTION:
All critically ill mechanically ventilated infants and children receive intravenous analgesic-sedatives which often include opiates and benzodiazepines (BENZO). Undesirable side effects from these drugs include respiratory depression, tolerance and dependence. Alpha 2-adrenergic receptor agonists, dexmedetomidine (DEX) and clonidine (CLON) have excellent sedative-analgesics effects, do not cause respiratory depression and are opiate/BENZO sparing. While both are efficacious in providing sedation, several factors have led to a substantial increase in the use of the newer drug DEX over the more established drug CLON in adults, children and infants. However, studies to guide therapy and dosing for infants and children are lacking. While these infants and children do require less opiate/BENZO therapy and fewer days on mechanical ventilation, they quickly develop tolerance to and have significant withdrawal from DEX. This necessitates protracted weaning of DEX and longer length of stay in the pediatric intensive care unit (PICU) since DEX can only be administered as a continuous intravenous (IV) infusion. CLON, on the other hand, has a longer half-life and has formulations that allow for continuous or intermittent IV and oral administration. Dr. Gauda has an approved IND to use the epidural formulation of CLON intravenously in infants and children. The purpose of this pilot study is to determine the effective IV dosing scheme of CLON that can be safely used as an adjunct to analgesic-sedation management for infants and children in the PICU. It will include a total of 24 infants and children with 4 CLON and DEX exposed in each age stratum: 0-3, 4-6, and 7-12 months. We hypothesize that IV CLON can achieve optimal sedation and reduce the need for opiate/BENZO therapy in critically ill infants and children who would otherwise receive DEX, and thus, reduce the length of stay in the PICU. Data from this study will be used to inform a larger randomized trial and will directly benefit infants and children in Baltimore who are critically ill. Funds are requested to cover the cost of the CLON drug levels and the investigational pharmacy.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children age: 0-12 months
* Intubated and mechanically ventilated in the JHH PICU
* Meet criteria for starting dexmedetomidine (per PICU protocol)

Exclusion Criteria:

* Postoperative from complex congenital heart disease
* Asphyxia
* Traumatic Brain Injury
* Major Chromosomal anomaly (Trisomy 13, 18)
* Any infant or child who is receiving ECMO therapy
* If death is considered imminent

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2015-09; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Sedation | 2-8 weeks
  Time spent (hrs) with a State Behavioral Scale <1 without the concurrent escalation of opiates or sedatives within 24 hrs after starting the CLON or DEX

SECONDARY OUTCOMES:
Frequency of cardiovascular occurrences | 2 - 8 weeks
  Frequency of cardiovascular occurrences i. ≥10 torr reduction in mean arterial blood pressure (MAP) ii. 20% drop in HR from the infant's baseline iii. Changes in HR or Blood pressure that triggers an intervention by the clinical team such as: -
  1. Adding or escalating cardiotonic meds
  2. holding the dose of timed sedative/analgesia
Length of stay | 2-8 weeks
  Length of stay in PICU for sedative-analgesic therapy after stabilization and extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Sapna R Kudchadkar, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States